CLINICAL TRIAL: NCT00113412
Title: A Multi-Center, Double-Blind, Randomized, Placebo-Controlled Study Of Orally Administered SP01A As Monotherapy Treatment Of HIV-Infected Patients
Brief Title: A Study of an Oral Entry Inhibitor, SP01A, in Treatment-Experienced HIV-Infected Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samaritan Pharmaceuticals, Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP01A-105-04
Record Dates: First submitted 2005-06-07; First posted 2005-06-08 (Estimated); Last update posted 2006-03-22 (Estimated); Status verified 2006-03

CONDITIONS: HIV Infections
Keywords: HIV; Treatment Experienced
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Drug: SP01A

SUMMARY:
One measurement of an HIV infected person's risk of progressing to AIDS is the number of viral particles of HIV in their blood (called a "viral load"). In a previous phase I/II study, SP01A was observed to significantly lower the amount of HIV in blood, improve quality of life (how well subject's felt), have a favorable safety profile (minimal side effects), and be well tolerated. Moreover, in in vitro testing SP01A: (1) demonstrated comparable or greater efficacy than currently approved anti-HIV drugs in preventing HIV virus replication; (2) was observed to have minimal toxic effect on human cells; and (3) demonstrated significant efficacy in preventing virus replication of HIV virus strains that resist currently approved anti-HIV treatments. Based on these results, SP01A demonstrates promise as a new and novel anti-HIV treatment.

The goal of this study is to further look at the dose response, efficacy, and safety of SP01A as monotherapy, given as a capsule to be swallowed, in the treatment of HIV-infected subjects. The investigators want to see if SP01A will lower the amount of HIV in blood.

Subjects will be assigned by chance to 1 of 4 groups. Neither the subject nor the study doctor or nurse will know which dose of the study drug the subject is taking or if the subject is receiving the placebo (a capsule that looks like the study drug but does not contain any active ingredient).

At the end of the 10-day study, the subject will be offered testing of their virus for resistance to approved drugs (genotype) and transferred to their physician for continued treatment with FDA-approved antiretroviral therapies. If the subject experiences a side effect, which continues past the end of the study, they will be further monitored until the side effect goes away.

DETAILED DESCRIPTION:
This is a multi-center, double-blind, randomized, placebo controlled Phase II study of orally administered SP01A as monotherapy treatment in HIV-infected patients with evidence of resistance to currently available antiretroviral therapy. This monotherapy study focuses on HIV-infected subjects who have previously failed antiretroviral regimens (treatment failures; defined as individuals with evidence of their viral load going up despite taking their anti-HIV drugs precisely as prescribed).

HIV-positive subjects will be evaluated during the pre-study period. Following a 4-week washout period (to ensure that any previous anti-HIV drug no longer remains in their system), all study groups will initiate the 10-day monotherapy study.

At the conclusion of the 10-day monotherapy study, subjects will have the option of having testing to determine the best anti-HIV treatment combination for their further treatment. Further treatment, if indicated, will be limited to FDA-approved anti-HIV treatments.

The primary objective of this study is to assess the dose-response, efficacy and safety of orally administered SP01A as monotherapy treatment (study drug alone) of HIV-infected subjects with evidence of resistance to currently available anti-HIV drug therapy.

The primary analysis is the reduction in viral load (log10) within each SP01A study arm as well as within the placebo arm as measured from the first day of drug administration (DAY-1 (Baseline)) to the last day of study drug administration (DAY-11 (Study-End)).

The secondary analysis is the reduction in viral load (log10) across SP01A active arms measured from DAY-1 (Baseline) to DAY-11 (Study-End).

The investigators may also test the HIV in each patient's blood to determine if one or more HIV strains exists that are resistant to currently approved anti-HIV drugs. This testing will be conducted at DAY-1 and Day-11. Additionally, the investigators may test to determine whether the virus develops resistance to the study drug on DAY-11.

Safety will be assessed at each visit by laboratory evaluations, physical examination and/or questioning for side effects. In the event of side effects, dosing of study drug may be stopped according to provisions outlined in the protocol.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion into this study, patients must fulfill the following criteria prior to the first day of study drug (i.e. Study Day-1) unless otherwise noted.

* Patient must be capable of giving informed consent. The principal investigator or study nurse will be responsible for obtaining written informed consent from potential patients prior to conducting any testing for the screening visit.
* 2. Patient is HIV-positive and has treatment-experienced virologic failure or documented resistance. Treatment-experienced virologic failure is defined as patients meeting the following criteria; (1) previous experience with antiretroviral therapy from at least two of the approved antiretroviral classes (i.e. treatment with a nucleoside reverse transcriptase inhibitor, and/or non-nucleoside reverse transcriptase inhibitor, and/or protease inhibitor) for three to six months; (2) increasing HIV RNA after treatment had previously lowered viral load to low or undetectable levels; (3) increasing viremia (HIV RNA > 5,000 copies/mL) in at least two viral load tests confirming their failing regimen. A patient does not need to currently be on therapy. A patient that is currently on a stable antiretroviral regimen that is successfully suppressing or maintaining viremia at low detectable levels (HIV RNA < 5,000 copies/mL) is not eligible for entry into the study.
* Patient has been off all anti-viral medications, including any unapproved or experimental treatment for HIV and antiretrovirals, for at least 4 weeks prior to Study Day-1 (baseline). The patient may initiate this 4 week period after screening, if, in the judgment of the principal investigator, the patient qualifies for the study.
* Patient is at least 18 years of age and not older than 60 years of age.
* Patient is capable of adhering to the protocol.
* Patient has a CD4+ count >50 cells/ml.
* Patient has a viral load of > 5000 copies/ml.
* Patient has a Karnofsky score greater than or equal to 60.
* Female patients that are of childbearing potential: (1) have a negative urine pregnancy test at screening, and agree to use a condom and another form of contraception from the start of the study; or (2) are incapable of becoming pregnant.

Exclusion Criteria:

Patients are ineligible to participate in the study if ANY of the following criteria are met.

* Patients with known or suspected allergy to procaine hydrochloride.
* Patients using sulfonamides (including Septra/Bactrim). Sulfonamides should not be used while on SP01A, because procaine will inactivate it. If a patient must be treated with Septra/Bactrim, that patient will be removed from the study.
* Patients with glaucoma using anti-cholinesterase inhibitors (Humorsol [demecarium bromide] echothiophate iodide, Floropryl [isoflurophate], Isopto-Eserine [physostigmine salicylate]). Anti-cholinesterase inhibitors should not be used while on SP01A, since anticholinesterases inhibit the breakdown of procaine hydrochloride.
* Patients with SGOT baseline value >3 times upper limit.
* Patients with SGPT baseline value >3 times upper limit.
* Patients with creatinine >2.0 mg/ dl.
* Patients with absolute neutrophil count <1,000 cells/mm3.
* Patients with platelets baseline value <75,000 cells/µl.
* Patients that currently have any active opportunistic infection. Prophylaxis for Mycobacterium avium intracellulare (MAI), cytomegalovirus (CMV), Pneumocystis carinii pneumonia (PCP), or herpes is permitted (excluding treatment with Sulfonamides).
* Females that are pregnant or breast feeding.
* Female patients of childbearing age who cannot either use dual contraception or abstain from sexual intercourse during the clinical study.
* Patients with less than 6 months life expectancy.
* Patients with active hepatitis (viral or drug induced).
* Patients with cancer, except peripheral (dermal) Kaposi's sarcoma.
* Patients on dialysis.
* Patients that currently have an active alcohol or substance abuse problem.
* Patients with any medical, psychological, psychiatric or substance use problem that, in the opinion of the principal investigator, will interfere with the patient's ability to complete the study.
* A patient that is currently on a stable antiretroviral regimen that is successfully suppressing or maintaining viremia at low detectable levels (HIV RNA < 5,000 copies/ml) is not eligible for entry into the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32
Dates: Start 2005-05

PRIMARY OUTCOMES:
The primary objective of this study is to assess the dose-response, efficacy, and safety of orally administered SP01A as monotherapy treatment in HIV-infected patients with evidence of resistance to currently available antiretroviral therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Erasto Saldi, MD, Study Director — Samaritan Pharmaceuticals, Inc
Locations (7):
- United States (7):
  - Therafirst Medical Centers, Fort Lauderdale, Florida
  - BioCollections Worldwide, Inc., Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Infectious Disease Research Institute, Tampa, Florida
  - Anderson Medical Group, Pittsburgh, Pennsylvania
  - Tarant County Infectious Disease, Fort Worth, Texas
  - University of Texas Health Science Center, Houston, Texas

REFERENCES:
- [Background] Xu J, Lecanu L, Han Z, Yao Z, Greeson J, Papadopoulos V. Inhibition of adrenal cortical steroid formation by procaine is mediated by reduction of the cAMP-induced 3-hydroxy-3-methylglutaryl-coenzyme A reductase messenger ribonucleic acid levels. J Pharmacol Exp Ther. 2003 Dec;307(3):1148-57. doi: 10.1124/jpet.103.055178. Epub 2003 Oct 14. PMID 14560037